CLINICAL TRIAL: NCT03589157
Title: Comparison of Safety and Efficacy of Coronary Drug-coated Balloon (DCB) Combined With Spot Stenting of Drug-eluting Stent (DES) Versus Second-generation DES for Treating Diffuse Coronary Artery Lesions: a Prospective, Randomized, Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-G-H-1518
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Diffuse Coronary Artery Lesions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon group (Experimental)
  Interventions: Device: drug-coated balloon (DCB) combined with spot stenting of drug-eluting stent (DES)
- second-generation drug-eluting stent group (Active Comparator)
  Interventions: Device: drug-coated balloon (DCB) combined with second-generation of drug-eluting stent (DES)

INTERVENTIONS:
Device: drug-coated balloon (DCB) combined with spot stenting of drug-eluting stent (DES) — using drug-coated balloon (DCB) combined with spot stenting of drug-eluting stent (DES) for treating diffuse coronary artery lesions
  Arms: Drug-coated balloon group
Device: drug-coated balloon (DCB) combined with second-generation of drug-eluting stent (DES) — using drug-coated balloon (DCB) combined with second-generation DES for treating diffuse coronary artery lesions
  Arms: second-generation drug-eluting stent group

SUMMARY:
The prospective, randomized, controlled clinical trial aims to evaluate the safety and efficacy of paclitaxel-eluting PTCA-balloon catheter (SeQuent® Please) combined with provisional spot stenting of DES versus DES for treating diffuse coronary artery lesions concerning interventional therapy and vessel patency.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related

  * Patients who have typical angina pectoris symptoms with obvious evidence of ischemia;
  * Patients whose ages are between 18-80 years;
  * Patients who must agree to receive a 9-month angiographic follow-up;
  * Patients who must agree to receive clinical follow-up of 30 days, and 3, 6, 9, 12, 24 and 36 months;
  * Patients who can understand the purpose of this study both psychologically and linguistically, demonstrating sufficient compliance to the study protocol;
  * Patients who express their recognition of the risks and benefits described in the informed consent form by providing their inform consent;
* Lesion-related

  * Diffuse coronary artery disease in situ;
  * Reference target vessel diameter of 2.5-4.0 mm and length of > 25 mm;
  * Non-target vessel lesions needing to receive a successful intervention therapy first before randomization to receive treatment for target lesions (note: within the same hospitalization);
  * Visually estimated diameter stenosis of ≥70%, or diameter stenosis of ≥50% with objective evidences of ischemia (treadmill exercise testing, ECT or FFR<0.8)

Exclusion Criteria:

* Patient-related:

  * Patients who have the attack of myocardial infarction within the past week, or whose troponin fails to return to normal although myocardial infarction has occurred for over one week;
  * Patients with serious congestive heart failure or NYHA IV-level serious heart failure;
  * Patients whose left ventricular ejection fraction is < 30%;
  * Patients who have medical history of stroke or TIA within 6 months prior to the surgery;
  * Patients who have a current or previous history of serious liver failure and thereby fail to meet the requirements of angiography;
  * Patients who have a current or previous history of serious kidney failure (GFR<30 ml/min) and thereby fail to meet the requirements of angiography;
  * Patients who have a previous history of intracranial neoplasms, aneurysm, arteriovenous malformation or cerebral hemorrhage;
  * Patients whose life expectancy does not exceed 1 year or who are difficult to follow up clinically;
  * Patients who have been scheduled to undergo elective surgery which may lead to the early discontinuation of ADP receptor antagonists;
  * Pregnant or lactating women or women who are planning to become pregnant during the study.
  * Patients participating in any other clinical trial;
  * Patients who are considered not suitable for inclusion by the investigator for any other reason;
* Lesion-related:

  * Patients who have the evidence of extensive thrombosis in target vessels prior to the interventional therapy;
  * Patients who have left main coronary artery disease or graft lesions needing to be treated;
  * Patients who have bifurcation lesions with a side-branch vessel diameter of >2.5 mm;
  * Patients who have lesions at the ostia of coronary artery, at the circumflex branch, at the ostia of anterior descending branch or within 5 mm at the ostia of coronary artery;
  * Severe intimal tear disease;
  * In-stent restenosis;
  * Lesions which can not be treated with PTCA or other intervention technologies;
  * Lesions with serious calcification;
* Concomitant medication related

  * Patients who have a physique prone to hemorrhage and are prohibited from taking anticoagulants or antiplatelet drugs;
  * Patients who can not tolerate Aspirin and/or Clopidogrel, or who have serious hypohepatia and must not use Clopidogrel;
  * Patients who can not tolerate or have known allergy to heparin, contrast media, paclitaxel, iopromide, rapamycin, poly(lactic-co-glycolic acid) polymers or stainless steel, etc,;
  * Patients with a history of leukopenia (with WBC<3×109/L for more than 3 days), neutropenia (with ANC <1,000 cells/mm3 for more than 3 days), or thrombocytopenia (with platelet count <100,000/mm3);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss | 9 months
  Late lumen loss (LLL) in the lesion segment within 9 months after surgery

SECONDARY OUTCOMES:
Interventional therapy success rate | 3 years
  including device success rate, lesion success rate and clinical success rate
Restenosis rate (RR) in the lesion segment | 9 months
  Restenosis rate (RR) in the lesion segment on 9 months after operation
Clinically-driven target lesion revascularization | 3 years
  Clinically-driven target lesion revascularization (CD-TLR) at 30 days and 3, 6, 9, 12, 24 and 36 months postoperatively
Device-related cardiovascular clinical composite endpoints | 3 years
  including cardiac death, target vessel myocardial infarction, and clinically-driven target lesion revascularization (CD-TLR), called target lesion failure (TLF) for short
Patient-related cardiovascular clinical composite endpoints | 3 years
  including all-cause mortality, all myocardial infarctions, and any revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — Chinese PLA General Hospital